CLINICAL TRIAL: NCT03044041
Title: Topical Intra-Articular High Doses Compared With Low Doses of Tranexamic Acid to Reduce Blood Loss in Primary Total Knee Arthroplasty: A Double-Blind Randomized Controlled Trial
Brief Title: Comparison Between Low Dose and High Dose Intra-articular Tranexamic Acid in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OrthoTU08
Record Dates: First submitted 2017-01-29; First posted 2017-02-06 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Blood Loss, Surgical
Keywords: Blood loss; Tranexamic acid; Total knee arthroplasty; Topical administration
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): single dose of intra-articular Tranexamic acid 500 miligrams
  Interventions: Drug: Tranexamic Acid
- High dose (Active Comparator): Single dose of intra-articular Tranexamic acid 3 grams
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — IA (intra-articular) tranexamic acid after capsule closure

SUMMARY:
The purpose of this study is to compare blood loss between using low dose (500 mg) and high dose (3 g) topical intra-articular tranexamic acid after total knee arthroplasty in double-blind RCT

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritic knee who underwent primary total knee arthroplasty

Exclusion Criteria:

* Abnormal coagulation or bleeding disorder
* Allergy to tranexamic acid
* History of thromboembolism or ischemic heart disease or cerebrovascular accident
* chronic kidney disease stage 3-4

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Total blood loss | 72 hours after TKA
  Blood loos that calculated from Haemoglobin drop at 72 hours after surgery

SECONDARY OUTCOMES:
Blood transfusion | 0-72 hours after surgery
  incidence of blood transfusion after surgery
Rate of participants with thromboembolism | At 72 hours and 2 weeks after surgery
  Clinical thromboembolism after surgery
Rate of participants with infection | 0-3 months after surgery
  Superficial or deep infection after TKA
Knee ROM | At 2, 6 weeks after surgery
  Range of motion of the knee
Functional score | At 6 weeks after surgery
  Modified WOMAC

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Klong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided